CLINICAL TRIAL: NCT04603040
Title: A Single-arm, Multicenter, Phase II Clinical Study to Evaluate the Efficacy and Safety of Toripalimab Injection (JS001) in the Treatment of Recurrent or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma Who Have Failed at Least Two Prior Lines of Therapy and Are Positive Specific Markers
Brief Title: A Study to Evaluate the Efficacy and Safety of Toripalimab Injection in the Treatment of Recurrent or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma Who Have Failed at Least Two Prior Lines of Therapy and Are Positive Specific Markers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001-033-II-GC
Record Dates: First submitted 2020-09-17; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-01

CONDITIONS: Recurrent or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma Who Have Failed at Least Two Prior Lines of Therapy
MeSH Terms: conditions — Recurrence | interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental group (Experimental): Experimental group:ToripalimabTreatment
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — Experimental group:
  Toripalimab, 240mg, IV infusion, every 3 weeks (q3w), In a cycle of 3 weeks (21 days), until occurrence of termination event specified in the protocol.
  Other Names: Tuoyi

SUMMARY:
This is a single-arm, multicenter, phase 2 study to assess the efficacy and safety of Toripalimab Injection (JS001) in patients with advanced recurrent or metastatic gastric or gastroesophageal junction adenocarcinoma who have failed at least 2 prior lines of therapy and are positive for specific markers.

Patients who meet the requirements will be treated with Toripalimab injection 240 mg once every 3 weeks (q3w) until disease progression based on imaging according to RECIST 1.1 criteria judged by the investigator, or intolerable toxicity, or withdrawal of informed consent, or withdrawal of treatment judged by the investigator, or voluntarydiscontinuation of treatment by the patient with CR of more than 6 months, or up to 2 years of treatment for JS001, whichever occurs first.

For the case that the patient shows disease progression on imaging according to RECIST 1.1, as long as the investigator judges that the patient can still benefit from continued medication, the treatment with Toripalimab Injection can be continued until the progression on imaging assessed by the investigator for the second time. The clinical benefit is based on the results of comprehensive assessment by the investigator in combination with imaging findings and clinical condition when the patient has no intolerable toxicity or the symptoms worsen due to disease progression.

Tumor assessments are performed at screening (as the baseline), every 6 weeks from the first dose in the first year, and every 9 weeks from the second year until radiologically documented progressive disease (PD), or second disease progression judged by the investigator (for patients with disease progression shown by first imaging, but who can continue treatment judged by the investigator), or withdrawal of informed consent by the patient, or loss to follow-up, or start of a new anti-tumor therapy, or the termination of the study. If a patient withdraws from the study for reasons other than disease progression (including due to the AE or because the treatment interval is beyond the window) and no disease progression occurs at the time of withdrawal, radiographic assessments should be continued until disease progression, death, or start of a new anti-tumor therapy. Patient medication management is based on the investigator's tumor assessment.

ELIGIBILITY:
1. Patients voluntarily participate in this study after full informed consent and sign a written informed consent form; 2. Age ≥18 years and ≤75 years at the time of signing informed consent; 3. Histologically or cytologically confirmed gastric or gastroesophageal junction adenocarcinoma; 4. Disease progression after at least two lines of previous treatment for recurrent or metastatic gastric or gastroesophageal junction adenocarcinoma:

1. First-line treatment must be combination regimen of two or more chemotherapy drugs and disease progression occurs; or distant metastasis or local recurrence within 6 months after completion of radical neoadjuvant chemotherapy or adjuvant chemotherapy (or chemoradiotherapy) based on platinum-based combination chemotherapy, which can be considered as progression after first-line treatment;
2. Second-line treatment includes but is not limited to chemotherapy, anti-angiogenic therapy and disease progression occurs;
3. Patients known to be HER2-positive require treatment with approved anti-HER2 targeted agents.
4. The interval between the end of systemic treatment and the first study drug administration is at least 4 weeks (the washout period of oral fluorouracil drugs is 2 weeks); 5. Previous tumor samples or fresh tumor tissue biopsy samples can be provided, and any of the following biomarkers are confirmed positive by the central laboratory:

1)PD-L1 positive: defined as PD-L1 staining positive at any intensity in ≥5% tumor cells (TC) or ≥10% immune cells (IC); 2)Epstein-Barr virus (EBV) positive: defined as positive for EBV-encoded small RNA in situ hybridization (EBER-ISH); 3)Tumor mutation burden-high (TMB-H): tumor tissues will be detected by whole exome sequencing (WES), with tumor mutation burden ≥12 Muts/Mb; 4)Microsatellite instability-high (MSI-H): Tumor tissue is tested by whole exome sequencing (WES) to confirm MSI-H positivity; 6. at least one measurable lesion according to RECIST 1.1 assessment criteria; 7. expected survival ≥3 months; 8. According to the Eastern Cooperative Oncology Group (ECOG) criteria (Section 11.2 Appendix 2), the performance status score is 0 or 1; 9. Good organ function:

1. Hematology (no blood transfusion or colony-stimulating factor and thrombopoietin 14 days before the first study drug administration) Neutrophil count≥1.5×109/L; Thrombocyte count≥100×109/L; Hemoglobin≥90 g/L;
2. Kidney function Serum creatinine≤1.5 x upper limit of normal (ULN) or Calculated creatinine clearance by referring to the Cockcroft-Gault formula (Section 11.6 Appendix 6) or site practice≥50 mL/min;
3. Hepatic function Bilirubin total≤1.5 x ULN or ≤3 x ULN (patients with known Gilbert's disease) ; ALT/AST≤3 x ULN (without liver metastasis) or ≤5 x ULN (in case of liver metastases) ; Alkaline phosphatase≤3 x ULN (without liver and bone metastasis) or ≤5 x ULN (in case of liver or bone metastasis) ; Albumin≥30 g/L;
4. Coagulation function:International normalized ratio (INR) or prothrombin time (PT) or activated partial thromboplastin time (aPTT) ≤1.5 x ULN.

10. Adverse events and/or complications caused by any previous treatment, including surgery or radiotherapy, have been fully relieved and must have been relieved to grade 0 or 1 [according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE 5.0)]; except for alopecia/pigmentation of any grade and long-term toxicity caused by other treatments, which cannot be recovered and does not affect the study drug administration/compliance and patient safety in the judgment of the investigator; 11. Within 7 days before the first dose, women of childbearing age must confirm that the serum pregnancy test is negative and agree to use effective contraceptive measures during the use of the study drug and within 60 days after last dose. A female of childbearing potential in this protocol is defined as a sexually mature female who:

1. No hysterectomy or bilateral oophorectomy,
2. Spontaneous menopause does not last for 24 consecutive months (amenorrhea after cancer treatment and not rule out fertility) (i.e., menstruation at any time within the previous 24 consecutive months).

Male patients with partners of childbearing potential must agree to use effective contraception during the use of the study drug and within 60 days after last dose.

Exclusion criteria:

1. With pathologically diagnosed squamous cell carcinoma or sarcoma or undifferentiated carcinoma of the stomach or gastroesophageal junction;
2. Patients with necrotic lesions, judged by the investigator to have a risk of massive hemorrhage;
3. Symptomatic spinal cord compression, or untreated patients expected to have symptoms of spinal cord compression; or for previously diagnosed and treated spinal cord compression, there is no evidence that the disease is clinically stable for ≥4 weeks before the first study drug administration; 1)Patients with asymptomatic spinal cord compression indicated by imaging, which is assessed as stable by specialists, unless treatment for spinal cord compression is not required temporarily;
4. Poorly controlled pleural effusion, pericardial effusion or ascites requiring regular drainage;
5. Accompanied by severe peritoneal metastasis, mainly manifested as: clinically significant intestinal obstruction; moderate to large amount of ascites; barium enema revealed small intestinal stenosis;
6. Poorly controlled tumor-related pain; 1)For patients requiring analgesics, treatment must be on a stable dose prior to study participation; 2)Symptomatic lesions suitable for palliative radiotherapy (e.g., bone metastasis or metastasis resulting in nerve injury) should be treated before enrollment; 3)Prior to enrollment, local treatment of asymptomatic metastatic lesions that may cause functional deficit or intractable pain due to further growth (e.g., current epidural metastases not associated with spinal cord compression) should be considered if appropriate;
7. Active or untreated CNS metastases as determined by computed tomography (CT) or magnetic resonance imaging (MRI) assessment during screening and previous imaging assessment; 1)Patients who have previously received treatment for CNS metastases, shown to be stable for ≥4 weeks by imaging examination during the screening period, and stopped systemic hormone therapy (prednisone or other hormones with equal efficacy at a dose > 10 mg/day) for ≥4 weeks before the first study drug administration can participate in the study;
8. Patients with a history of carcinomatous meningitis;
9. Patients with a weight loss of more than 10% within 2 months before signing the informed consent form;

   Exclusion criteria for concurrent other diseases or concomitant conditions:
10. Patients with other malignant tumors except for gastric cancer (except for cured cervical carcinoma in situ, basal or squamous cell skin cancer, localized prostate cancer with radical treatment, ductal carcinoma in situ with radical treatment) within 5 years before the first study drug administration;
11. Within 28 days prior to the first study drug administration, there are other major surgeries except for the diagnosis of gastric cancer, or major surgeries are expected to be performed during the study, unless assessed by researchers and specialists that they have fully recovered from the complications of major surgery;
12. Clinically significant underlying medical conditions (e.g., dyspnea, pneumonia, pancreatitis, poorly controlled diabetes, active or poorly controlled infection, drug or alcohol abuse, or psychiatric disorders) that, in the opinion of the investigator, can affect study drug administration and protocol compliance;
13. Presence of severe neurological or psychiatric disorders, including dementia and epileptic seizures;
14. Have NCI-CTCAE ≥grade 2 peripheral neuropathy;
15. Pregnant or lactating female patients;
16. Patients with major cardiovascular diseases, such as heart disease of New York Heart Association (NYHA) functional class II or above (see Section 11.5 Appendix 5), myocardial infarction within 3 months before the first study drug administration, poorly controlled arrhythmia or unstable angina;

1)Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction < 50% must be treated with an optimized stable medical regimen at the discretion of the treating physician, with consultation with a cardiologist, as appropriate;

Exclusion criteria for medication:

17. Previous history of hypersensitivity to other monoclonal antibodies or any component of Toripalimab Injection (JS001); 18. Previous treatment targeting PD-1 receptor or its ligand PD-L1 or cytotoxic T-lymphocyte-associated protein 4 (CTLA4) receptor; 19. Participated in or planned to participate in other intervention studies within 4 weeks before the first study drug administration.

20. Treatment with systemic immunostimulatory drugs (including but not limited to interferon or IL-2) within 2 weeks or 5 half-lives of the drug (whichever is longer) before the first study drug administration; 21. Received systemic corticosteroids (> 10 mg/day prednisone equivalent drug) or other systemic immunosuppressive agents (including but not limited to cyclophosphamide, azathioprine, methotrexate, thalidomide and anti-tumor necrosis factor drugs [anti-TNF]) within 2 weeks before the first study drug administration ;

1. Topical, ocular, intra-articular, intranasal, and inhaled corticosteroids are permitted;
2. Patients receiving acute low-dose systemic immunosuppressive agents (e.g., a single dose of dexamethasone for nausea) can be enrolled after discussion with and approval by the medical monitor;
3. Patients who need baseline and follow-up MRI/CT tumor assessment can use steroids prophylaxis if they have previous allergic reactions to intravenous contrast media.
4. Inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (e.g., fludrocortisone) for orthostatic hypotension, and low-dose corticosteroids for maintenance treatment of adrenocortical insufficiency are permitted;

Exclusion criteria for special immune status:

22. History of autoimmune diseases, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis (see Section 11.7, Appendix 7 for a more comprehensive list of autoimmune diseases);

1. Patients with autoimmune-related hypothyroidism on stable doses of thyroid hormone replacement are eligible for this study;
2. Patients with type 1 diabetes controlled on a stable insulin regimen are eligible for this study; 23. Patients with previous allogeneic bone marrow transplantation or previous solid organ transplantation; 24. Any live vaccine (e.g., vaccines against infectious diseases, such as influenza vaccine, varicella vaccine, etc.) within 4 weeks (28 days) before the first study drug administration; 25. Active infection, including tuberculosis (clinical diagnosis including clinical history, physical examination and imaging findings, as well as TB tests according to local medical routine), hepatitis B, hepatitis C or human immunodeficiency virus (HIV antibody positive);

1)Patients who are positive for hepatitis B surface antigen (HBsAg+) and/or hepatitis B core antibody (HBcAb+) are required to undergo hepatitis B virus deoxyribonucleic acid (HBV DNA) test. If HBV DNA copy number is ˂1000 cps/mL, or less than the lower limit of detectable value at the study site, the patients can participate in this study; 2)Patients who are positive for hepatitis C antibody (HCV Ab+) are required to have an HCV RNA test and are eligible for this study only if they are negative for HCV RNA (defined as below the lower limit of detectable value at the study site); 26. History of idiopathic pulmonary fibrosis, drug-induced pneumonia, organized pneumonia (i.e., bronchiolitis obliterans), idiopathic pneumonia, or evidence of active pneumonia on chest CT scan at screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 12 months
  ORR assessed by IRC according to RECIST v1.1 assessment criteria. ORR is defined as the proportion of subjects with best response of complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 12 months
  ORR assessed by the investigator according to RECIST v1.1 assessment criteria. ORR is defined as the proportion of subjects with best response of CR or PR.
DoR | Up to 12 months
  DoR is defined as the time from the first documented response until the first documented evidence of disease progression or death from any cause, whichever occurs first;
DCR | Up to 12 months
  DCR is defined as the proportion of patients with best response of CR or PR or stable disease (SD);
PFS | Up to 12 months
  PFS is defined as the time from enrollment to the first documentation of disease progression or death from any cause, whichever occurs first;
iORR | Up to 12 months
  iORR is defined as the proportion of subjects with best response of CR or PR;
iDoR | Up to 12 months
  iDoR is the time from the first documented response until the first documented evidence of disease progression or death from any cause, whichever occurs first;
iDCR | Up to 12 months
  iDCR is the proportion of patients with best response of CR or PR or SD;
IPFS | Up to 12 months
  IPFS is defined as the time from enrollment to the first documentation of disease progression or death from any cause, whichever occurs first;
Overall survival (OS) | Up to 12 months
  Overall survival (OS), defined as the time from enrollment to death of the patient from any cause.
PFS rates at 6 and 12 months | Up to 12 months
  It is defined as the proportion of patients alive without documented disease progression at 6 and 12 months after enrollment assessed by RECIST v1.1 criteria
OS rates at 9 months and 12 months | Up to 12 months
  defined as the proportion of patients alive at 9 months and 12 months after enrollment.

OTHER OUTCOMES:
Incidence of AEs/SAEs as Assessed by CTCAE v5.0 | Up to 12 months
  Analysis of adverse events (AEs) are based on treatment-related AEs (trAEs) and immune-related AEs (irAEs), and all-grade AEs and grade 3-4 AEs. AEs are evaluated by investigators according to the Common Terminology Criteria for Adverse Events, version 5.0
JS001 anti-drug antibody assessment | Up to 12 months
  Serum levels of Anti-drug antibody of JS001 treatment
Epidemiological data survey | Up to 12 months
  based on the patient data screened by this project, the proportion of PD-L1-positive, EBV-positive, TMB-H and MSI-H patients is assessed
JS001 anti-drug antibody assessment | Up to 12 months
  Incidence of Anti-drug antibody of JS001 treatment

CONTACTS AND LOCATIONS:
Locations (39):
- China (39):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Affiliated Hospital of Hebei University, Baoding
  - Peking University International Hospital, Beijing
  - Sichuan Cancer Hospital, Chengdu
  - The First Hospital of Jilin University, Ch’ang-ch’un
  - Fujian Provincial Cancer Hospital, Fuzhou
  - Union Hospital affiliated to Fujian Medical University, Fuzhou
  - Affiliated Tumor Hospital of Guangzhou Medical University, Guangzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - The sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - The First Affiliated Hospital of Zhejiang University Medical College, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Zhejiang University School of Medicine, Sir Run Run Shaw Hospital, Hangzhou
  - Affiliated Tumor Hospital of Harbin Medical University, Harbin
  - Anhui Provincial Hospital, Hefei
  - Second Affiliated Hospital of Anhui Medical University, Hefei
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - The First Affiliated Hospital of Bengbu Medical College, Hefei
  - Henan Cancer Hospital, Henan
  - The First Affiliated Hospital of Nanhua University, Hengyang
  - Shandong Cancer Hospital, Jinan
  - The first Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - Jiangxi Provincial Cancer Hospital, Nanchang
  - The First Affiliated Hospital of Nanchang University Junhe Li, Nanchang
  - Jiangsu Cancer Hospital, Nanjing
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - Nantong Tumor Hospital, Nantong
  - Affiliated Hospital of Qingdao University, Qingdao
  - Shengjing Hospital of China Medical University, Shenyang
  - The First Affiliated Hospital of Soochow University, Suzhou
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - Shanxi Cancer Hospital, Taiyuan
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - The First Affiliated Hospital of Xinjiang Medical University, Xinjiang
  - Xuzhou Central Hospital, Xuzhou
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Zhengzhou Central Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No